CLINICAL TRIAL: NCT05814692
Title: Feasibility of BIOchemical Urine Analysis of Adherence to Statins and Associated FACTorS in Coronary Artery Disease: The BIO-FACTS Pilot Study
Brief Title: BIOchemical Urine Analysis of Adherence to Statins and Associated FACTorS in Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: BIO-FACTS
Record Dates: First submitted 2023-03-17; First posted 2023-04-18 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Coronary Heart Disease
Keywords: coronary artery disease; statin; atorvastatin; Rosuvastatin; adherence; biochemical urine testing of adherebnce
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — prospectively defined blood and urine sampling protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood and urine samples — blood and urine samples

SUMMARY:
Feasibilty study of biochemical urine analysis of adherence to high intensity statin therapy in outpatients with coronary artery disease

DETAILED DESCRIPTION:
Background:

Statin therapy is known to improve clinical outcomes in patients with coronary artery disease (CAD), while being highly cost-effective. However, adherence to statin therapy in real world settings is suboptimal and represents a possible target to ameliorate secondary CAD disease prevention. Previous interventional studies on statin adherence showed inconsistent results and it is widely acknowledged that a tailored adherence improvement approach adapted to patient determinants is required. However, methodology to accurately detect and characterize non-adherent patients is challenging and constitutes an important obstacle to developing such interventions. Urine analysis with liquid chromatography/mass spectrometry (LC-MS) for detection of statin intake is a promising method for objective measurement of adherence as an adjunct to subjective adherence assessment using questionnaires, which has not been applied in CAD patients in Germany.

Objectives: In this pilot study (i) a feasibility testing of objective (LC-MS urine analysis) and subjective (questionnaire survey) measures of adherence to statin therapy will be performed, (ii) the prevalence of nonadherence in the target population will be determined , and (iii) instruments assessing possible factors associated with (non-)adherence (e.g. side effects, beliefs about medications, and disease-related knowledge) will be evaulated, in order to establish a methodological ground for further studies characterizing non-adherent patients.

Methods:

Outpatients with CAD treated in University Hospital Düsseldorf and receiving guideline-recommended atorvastatin or rosuvastatin on prescription will be included in the pilot study. Based on sample size calculation about 130 patients will be recruited. A biochemical method of objective urine measurement of statin intake by LC-MS will be combined with a preselected set of questionnaires on adherence behavior and associated factors. Clinical characteristics will be obtained from patient records. A sub-sample of the study population will be invited to participate in the interview for the evaluation of the questionnaire survey.

Outlook:

Based on the results of the pilot study, an adequately powered study to characterize non-adherent patients and identify patterns of non-adherence will be conducted. The results will be used for the development of a complex tailored intervention for non-adherent patients in Germany.

ELIGIBILITY:
Inclusion Criteria:

* patients with coronary artery disease
* prescription of atorvastatin or rosuvastatin

Exclusion Criteria:

* < 18 years
* impairment (e.g. dementia)
* language barrier (German)
* end-stage kidney disease with hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with coronary artery disease and prescription of atorvastatin or rosuvastin
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Recrutiment Rate | through study completion, approximately 1 year
  Recruitment will be assessed by proportion of eligible patients (in %) that agree to participate in the study
Rate of participating patients (in %) from whom a urine sample can be obtained that is suitable for detection analysis of atorvastatin or rosuvastatin by liquid chromatography/mass spectrometr | through study completion, approximately 1 year
  Rate of participating patients (in %) from whom a urine sample can be obtained that is suitable for detection analysis of atorvastatin or rosuvastatin by liquid chromatography/mass spectrometry
Rate of urine samples (in %) from which a valid result of liquid chromatography/mass spectrometry analysis for detection of atorvastatin or rosuvastatin can be obtained. | through study completion, approximately 1 year
  Rate of urine samples (in %) from which a valid result of liquid chromatography/mass spectrometry analysis for detection of atorvastatin or rosuvastatin can be obtained.
Average time (in minutes) that is needed by the study personnel to inform the patient about the study, receive written informed consent, hand out and retrieve the study questionnaire, and obtain a urine sample from the participant. | through study completion, approximately 1 year
  Average time (in minutes) that is needed by the study personnel to inform the patient about the study, receive written informed consent, hand out and retrieve the study questionnaire, and obtain a urine sample from the participant.
Average time (in minutes) that is needed by the participants to complete the study questionnaire | through study completion, approximately 1 year
  Average time (in minutes) that is needed by the participants to complete the study questionnaire
Rate of questions (in %) in the study questionnaire that are completely answered by participants | through study completion, approximately 1 year
  Rate of questions (in %) in the study questionnaire that are completely answered by participants

SECONDARY OUTCOMES:
Rate of patients (in %) in whom atorvastatin or rosuvastatin is detected by liquid chromatography/mass spectrometry analysis of a urine sample | through study completion, approximately 1 year
  Prevalence of statin adherence assessed by urine analysis
Rate of patients (in %) who report good adherence atorvastatin or rosuvastatin assessed by Medical Adherence Report Scale (MARS-D) | through study completion, approximately 1 year
  Prevalence of statin adherence assessed by questionnaire
Rate of patients (in %) from whom information on concomitant medication other than atorvastatin or rosuvastatin can be obtained from medical records | through study completion, approximately 1 year
Rate of patients (in %) from whom information on comorbidities (i.e., cerebrovascular disease, peripheral artery disease, arterial hypertension, and heart failure, or other comorbidities) can be obtained from medical records | through study completion, approximately 1 year
Rate of patients (in %) from whom socio-demographic information (i.e., level of education and income) can be obtained by the study questionnaire. | through study completion, approximately 1 year
  Rate of patients (in %) from whom socio-demographic information (i.e., level of education and income) can be obtained by the study questionnaire.
Rate of patients (in %) from whom information on perceived side-effects of statin therapy can be obtained by the study questionnaire (open question). | through study completion, approximately 1 year
  Rate of patients (in %) from whom information on perceived side-effects of statin therapy can be obtained by the study questionnaire (open question).
Rate of patients (in %) from whom information on patients' concerns about medications assessed by Beliefs about Medicines Questionnaire (BMQ-D) can be obtained by the study questionnaire | through study completion, approximately 1 year
  Rate of patients (in %) from whom information on patients' concerns about medications assessed by Beliefs about Medicines Questionnaire (BMQ-D) can be obtained by the study questionnaire
Rate of patients (in %) from whom information on anxiety and depression on the Hospital Anxiety and Depression Scale can be obtained by the study questionnaire. | through study completion, approximately 1 year
  Rate of patients (in %) from whom information on anxiety and depression on the Hospital Anxiety and Depression Scale can be obtained by the study questionnaire.
Rate of patients (in %) from whom information on health-related quality of life measured by the The Short Form (12) Health Survey (SF-12) can be obtained by the study questionnaire | through study completion, approximately 1 year
  Rate of patients (in %) from whom information on health-related quality of life measured by the The Short Form (12) Health Survey (SF-12) can be obtained by the study questionnaire
Rate of patients (in %) from whom information on social integration measured by the Social Integration Index can be obtained by the study questionnaire | through study completion, approximately 1 year
  Rate of patients (in %) from whom information on social integration measured by the Social Integration Index can be obtained by the study questionnaire
Rate of patients (in %) from whom information on social support measured by the Oslo-3-Social-Support-Scale can be obtained by the study questionnaire | through study completion, approximately 1 year
  Rate of patients (in %) from whom information on social support measured by the Oslo-3-Social-Support-Scale can be obtained by the study questionnaire
Rate of patients (in %) from whom information on health locus of control (open question) can be obtained by the study questionnaire | through study completion, approximately 1 year
  Rate of patients (in %) from whom information on health locus of control (open question) can be obtained by the study questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, Prof., Study Chair — Clinic for Cardiology, Pneumology and Angiology at University Hospital Düsseldorf
Locations (1):
- University-Hospital Düsseldorf Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No